CLINICAL TRIAL: NCT04713293
Title: China Pituitary Disease Registry Study
Brief Title: China Pituitary Disease Registry (CAPASITY)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, PhD, MD, Head of Department of Endocrine and Metabolism, Shanghai Jiaotong University School of Medicine, Chinese National Clinical Research Center for Endocrine and Metabolic Diseases (Shanghai), Shanghai Jiao Tong University School of Medicine
Other Study IDs: 1.0/20200606
Record Dates: First submitted 2020-12-31; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pituitary Disease
Keywords: Pituitary Disease; Pituitary Adenoma
MeSH Terms: conditions — Pituitary Diseases; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiologic studies have revealed a tremendous increase in the prevalence of pituitary disease and related mortality worldwide. In order to meet all the challenges in the treatment of pituitary disease in China, CAPASITY was founded in 2020. The objective of CAPASITY is to launch a pituitary disease management model based on the Internet health information platform. It allows the application and evaluation of pituitary disease treatment strategies at multiple centers. The proprietary electronic medical database will help the dynamic big-data analysis in epidemiology of pituitary disease, diagnosis, and treatment.

DETAILED DESCRIPTION:
In order to meet all the challenges in the diagnosis and treatment of pituitary diseases in China, CAPASITY was founded in 2020. With advanced medical equipment and Internet of Things (IoT) technology, CAPASITY is committed to creating an online and offline integrated solution for pituitary disease, and for the entire spectrum of pituitary disease, to achieve a more convenient and precise model of care for patients. aiming to establish a platform with diagnosis and treatment of pituitary disease and their long-term follow-up. It allows the application and evaluation of treatment strategies at these centers.

Objective:

* The purpose of the present study is to establish a multi-center nationwide prospective database of patients with pituitary adenomas to explore the epidemiology, biochemical, and clinical outcome related to pituitary tumors and its complications, as well as other pituitary disease.
* To collect cross-sectional data from patients seen and treated at each center so as to evaluate: the current status of care of patients with pituitary disease and its related complications, as well as other risk factors treatment strategies at multiple centers.
* To collect the prospective data of patients treated at each center in order to evaluate the strategies for the achievement of treatment goals, changes in management, control of risk factors, incidence and progression of related clinical endpoints (including mortality), behavioral changes, as well as QoL.

Methods: After obtaining informed consent, patients will be invited and initiated with a comprehensive baseline evaluation at each CAPASITY center. Then patients will be followed by clinical/laboratory visits on according to individualized patient's treatment plans. A repeated comprehensive clinical and laboratory assessment for hormones and imaging, as well as complications will be scheduled once a year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years
* Patients diagnosed with pituitary adenomas, and other pituitary diseases
* Pituitary adenomas resected by transsphenoidal surgery were identified by histological diagnoses.
* Gender: males and females
* Provide written informed consent
* Satisfactory compliance

Exclusion Criteria:

* Patients with significantly reduced life expectancy (less than 2 years)
* With Drug abuse
* With AIDS or syphilis or infectious diseases such as viral tuberculosis in active phase at enrollment

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pituitary disease
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of functional pituitary adenoma | through study completion, an average of 1 year
  percentage of PRLoma, GHoma, ACTHoma, and etc
remission and recurrence rate of pituitary surgery | through study completion, an average of 1 year
  treatment outcome of pituitary adenoma. Results will be dichotomized as remission, persistence or recurrence.

SECONDARY OUTCOMES:
concentration of GH | through study completion, an average of 1 year
  changes in GH
concentration of IGF-1 | through study completion, an average of 1 year
  changes in IGF-1
concentration of PRL | through study completion, an average of 1 year
  changes in PRL
concentration of ACTH | through study completion, an average of 1 year
  changes in ACTH
concentration of cortisol | through study completion, an average of 1 year
  changes in cortisol
concentration of fT3 | through study completion, an average of 1 year
  changes in fT3
concentration of fT4 | through study completion, an average of 1 year
  changes in fT4
concentration of TSH | through study completion, an average of 1 year
  changes in TSH
pituitary MRI | through study completion, an average of 1 year
  changes in MRI of sellar area
percentage of hypopituitarism | through study completion, an average of 1 year
  percentage of hypopituitarism
percentage of diabetes insipidus, etc | through study completion, an average of 1 year
  percentage of diabetes insipidus, etc

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, MD, PHD, Principal Investigator — National Metabolic Management center (Shanghai)
Locations (1):
- National Metabolic Management center, Shanghai, Shanghai Municipality, China